CLINICAL TRIAL: NCT02456207
Title: A Phase II, Multi-center, Randomized and Open Study to Evaluate and Compare the PK, PD and Safety of SCT400 With Rituximab in Patients With CD20+ B-cell Non-Hodgkin's Lymphoma
Brief Title: A Pharmacokinetic Study Comparing SCT400 And Rituximab in Patients With B-cell Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCT400NHL2
Record Dates: First submitted 2015-05-24; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2014-05

CONDITIONS: B-cell Non Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): SCT400:375 mg/m2, iv, one infusion
  Interventions: Drug: SCT400
- Active Comparator (Active Comparator): Rituximab: 375 mg/m2, iv, one infusion
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: SCT400
  Arms: Experimental
Drug: Rituximab
  Arms: Active Comparator

SUMMARY:
The primary objective of the study is to assess the pharmacokinetic (PK) similarity of SCT400 versus rituximab (MabThera®) in patients with CD20+ B-cell Non-Hodgkin's Lymphoma.

The secondary objective of the study is to evaluate the pharmacodynamics (PD) and safety of SCT400 versus rituximab (MabThera®), as well as the presence of human anti-chimeric antibodies (HACA).

ELIGIBILITY:
Inclusion Criteria:

1. aged from 18 to 75 years;
2. having histologically confirmed NHL expressing CD20 antigen;
3. having obtained CR (complete remission) or CRu (uncertain complete remisson) after the prior therapy;
4. ECOG performance status of 0 to 1
5. expected survival of at least ≥ 3 months;
6. signed an informed consent form which was approved by the institutional review board of the respective medical center .

Exclusion Criteria:

1. had received rituximab or other anti-CD20(+) monoclonal antibody treatment within 1 year before enrollment;
2. having to be at least 4 weeks beyond prior anticancer therapy including corticosteroid, or have not recovered from significant toxicities of prior therapy;
3. participating in other clinical trial within 30 days before enrolment;
4. with serious hematologic dysfunction (white blood cell count of <3.0×103/uL; absolute neutrophil count of <1.5×103/ uL; platelet count of < 75×103/uL; hemoglobin level of < 8.0 g/dL); hepatic dysfunction (total bilirubin level of > 1.5×ULN; aspartate amino transferase (AST) and alanine amino transferase (ALT) levels of >2.5 × ULN; renal dysfunction (serum creatinine level of > 1.5×ULN ); and International normalized ratio (INR) and partial thromboplastin time or activated partial thromboplastin time (aPTT) > 1.5 × ULN (unless on therapeutic coagulation);
5. had received live vaccine within 4 weeks prior to study entry;
6. with other malignancies ; or central nervous system (CNS) lymphoma, AIDS-related lymphoma; or active opportunistic infection, a serious nonmalignant disease;
7. seropositive for HCV antibody, or HIV antibody, or hepatitis B virus surface antigen (HBsAg). HBc antibody seropositive, but HBV DNA and HBsAg negative patients may participle following consultation with a hepatitis expert regarding monitoring and use of HBV antiviral therapy, and provided they agree to receive treatment as indicated,
8. recent major surgery (within 28 days prior to study entry );
9. with a history of allergic reaction or protein product allergy including murine proteins;
10. pregnant or lactating or not accepted birth control methods including male patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) for SCT400 and rituximab concentrations | 85 days

SECONDARY OUTCOMES:
AUC for SCT400 and rituximab concentrations | 1 week ,2 weeks, 4 weeks, 8 weeks and 12 weeks
Maximum observed concentration of the SCT400 and rituximab | 85 days
Change from baseline of CD19+ , CD20+ B-cells | 85 days
Comparison of AEs between the two study arms | 85 days
Comparison of HACA between the two study arms | 85 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China